CLINICAL TRIAL: NCT03898947
Title: Evaluation of Endometrial Changes in Breast Cancer Women With or Without Hormonal Therapies
Brief Title: Endometrial Changes in Breast Cancer Women With or Without Hormonal Therapies
Acronym: BETA-1
Status: Completed | Type: Observational
Sponsor: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Antonio Simone Laganà, Principal Investigator, Università degli Studi dell'Insubria
Other Study IDs: BETA-1
Record Dates: First submitted 2019-03-30; First posted 2019-04-02 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Breast Cancer; Endometrial Cancer
Keywords: Tamoxifen; Aromatase inhibitors; Breast cancer; Endometrial cancer; Endometrial pathologies
MeSH Terms: conditions — Breast Neoplasms; Endometrial Neoplasms | interventions — Hysteroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Tamoxifen users: Women undergoing therapy with Tamoxifen after surgery for breast cancer.
  Interventions: Procedure: Diagnostic hysteroscopy and targeted endometrial biopsy
- Aromatase inhibitors: Women undergoing therapy with Aromatase Inhibitors after surgery for breast cancer.
  Interventions: Procedure: Diagnostic hysteroscopy and targeted endometrial biopsy
- No treatment: Women who did not undergo any hormonal therapy after surgery for breast cancer.
  Interventions: Procedure: Diagnostic hysteroscopy and targeted endometrial biopsy

INTERVENTIONS:
Procedure: Diagnostic hysteroscopy and targeted endometrial biopsy — Diagnostic hysteroscopy and targeted endometrial biopsy

SUMMARY:
A history of breast cancer is a risk factor for the development of endometrial pathologies, such as typical and atypical glandular hyperplasia, endometrial polyps, uterine fibroids, endometrial adenocarcinoma and uterine sarcoma, probably due to some common risk factors (eg. obesity, nulliparity). Even if ethiopathogenesis for breast cancer and endometrial pathologies is not well established, both genetic factors and hyperestrogenic state may be play a pivotal role for their development. Indeed, relative hyperestrogenism is also the main target for the treatment of breast cancer. Currently used therapies for this purpose are selective estrogen receptor (ER) modulators (SERMs), such as Tamoxifen (TAM), and third generation non-steroidal aromatase inhibitors (AIs), such as letrozole and anastrozole.

TAM has both agonist and antagonist properties, depending upon the individual target organ and circulating levels of serum estrogens: on the one hand, it blocks estrogen stimulation in breast tissue; on the other hand, TAM shows an ER agonist activity in the endometrium that is able to stimulate proliferation and, in some cases, it causes an increased risk of uterine pathologies. Women with hormone-dependent breast cancer have to use TAM for five to ten years. Many reports suggest that the risk of uterine pathologies increases with the time of administration.

Considering these elements, the primary aim of this study will be to investigate the incidence of endometrial pathologies, especially of endometrial cancer, in different groups of breast cancer women undergoing diagnostic hysteroscopy.

ELIGIBILITY:
Inclusion Criteria:

* History of breast cancer treated with surgery (regardless of the adjuvant radio/chemotherapy)

Exclusion Criteria:

* Incomplete data collection
* Recurrence of breast cancer
* Any other concomitant disease
* Any pharmacological treatment (wash-out: 3 months) other than Tamoxifen or Aromatase inhibitors
* Women who switched from a therapy to another one during the study period.

Ages: 18 Years to 80 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Breast cancer women with or without hormonal therapy, undergoing diagnostic hysteroscopy and targeted endometrial biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 1329 (Actual)
Dates: Start 2007-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Endometrial pathologies | 5 years after breast cancer surgery
  Rate of endometrial pathologies (benign or malignant)

CONTACTS AND LOCATIONS:
Overall Officials: Benito Chiofalo, M.D., Principal Investigator — "Regina Elena" National Cancer Institute of Rome

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chiofalo B, Mazzon I, Di Angelo Antonio S, Amadore D, Vizza E, Lagana AS, Vocaturo G, Calagna G, Favilli A, Palmara V, Maranto M, Vitale SG, Cucinella G, Granese R, Ghezzi F, Sperduti I, Triolo O. Hysteroscopic Evaluation of Endometrial Changes in Breast Cancer Women with or without Hormone Therapies: Results from a Large Multicenter Cohort Study. J Minim Invasive Gynecol. 2020 May-Jun;27(4):832-839. doi: 10.1016/j.jmig.2019.08.007. Epub 2019 Aug 16. PMID 31425735